CLINICAL TRIAL: NCT00863798
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study To Evaluate The Efficacy And Safety Of 2 Fixed Doses (10 And 50 mg/Day) Of DVS SR Tablets In Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release In Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3151A1-3362; B2061005; 3151A1-3362-US
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desvenlafaxine succinate sustained release 10 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release 10mg
- Desvenlafaxine succinate sustained release 50 mg (Experimental)
  Interventions: Drug: Desvenlafaxine Succinate Sustained-Release 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Desvenlafaxine Succinate Sustained-Release 10mg — 10 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained release 10 mg
Drug: Desvenlafaxine Succinate Sustained-Release 50 mg — 50 mg tablet, once daily dosing for 8 weeks
  Arms: Desvenlafaxine succinate sustained release 50 mg
Drug: placebo — Matching placebo tablets (10 or 50mg). Daily dosing for 10 +/- 4 days during a placebo lead-in period, and then 8 weeks during the double-blind period.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the antidepressant efficacy and safety of two doses of desvenlafaxine succinate sustained release (10 and 50 mg/day) in adults with Major Depressive Disorder. The study will also assess changes in sexual function and general and functional quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult, outpatient with primary diagnosis of Major Depressive Disorder (depressive symptoms for at least 30 days prior to screening).
* Hamilton Psychiatric Rating Scale for Depression (HAM-D 17) total score of >= 20.
* Clinical Global Impressions Scale-Severity (CGI-S) score of >= 4.

Exclusion Criteria:

* Clinical instability (25% or greater increase/decrease in HAM-D 17 total score from screening to baseline).
* Significant risk of suicide as assessed by clinician judgment, HAM-D 17 and Columbia Suicide-Severity Rating Scale scores Other eligibility criteria also apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (24):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Cromwell, Connecticut
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Salem, Oregon
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Herndon, Virginia
  - Pfizer Investigational Site, Midlothian, Virginia
  - Pfizer Investigational Site, Middleton, Wisconsin
  - Pfizer Investigational Site, Waukesha, Wisconsin

REFERENCES:
- [Derived] Zilcha-Mano S, Wang X, Wajsbrot DB, Boucher M, Fine SA, Rutherford BR. Trajectories of Function and Symptom Change in Desvenlafaxine Clinical Trials: Toward Personalized Treatment for Depression. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):579-584. doi: 10.1097/JCP.0000000000001435. PMID 34183490
- [Derived] Soares CN, Zhang M, Boucher M. Categorical improvement in functional impairment in depressed patients treated with desvenlafaxine. CNS Spectr. 2019 Jun;24(3):322-332. doi: 10.1017/S1092852917000633. Epub 2017 Nov 15. PMID 29140227
- [Derived] McIntyre RS, Fayyad R, Mackell JA, Boucher M. Effect of metabolic syndrome and thyroid hormone on efficacy of desvenlafaxine 50 and 100 mg/d in major depressive disorder. Curr Med Res Opin. 2016;32(3):587-99. doi: 10.1185/03007995.2015.1136603. Epub 2016 Jan 13. PMID 26709542
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. A Post Hoc Analysis of the Effect of Weight on Efficacy in Depressed Patients Treated With Desvenlafaxine 50 mg/d and 100 mg/d. Prim Care Companion CNS Disord. 2015 Jun 4;17(3):10.4088/PCC.14m01741. doi: 10.4088/PCC.14m01741. eCollection 2015. PMID 26644956
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058
- [Derived] Soares CN, Endicott J, Boucher M, Fayyad RS, Guico-Pabia CJ. Predictors of functional response and remission with desvenlafaxine 50 mg/d in patients with major depressive disorder. CNS Spectr. 2014 Dec;19(6):519-27. doi: 10.1017/S1092852914000066. Epub 2014 Feb 26. PMID 24571916
- [Derived] Liebowitz MR, Tourian KA, Hwang E, Mele L; Study 3362 Investigators. A double-blind, randomized, placebo-controlled study assessing the efficacy and tolerability of desvenlafaxine 10 and 50 mg/day in adult outpatients with major depressive disorder. BMC Psychiatry. 2013 Mar 22;13:94. doi: 10.1186/1471-244X-13-94. PMID 23517291
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3151A1-3362&StudyName=Study%20Evaluating%20Desvenlafaxine%20Succinate%20Sustained%20Release%20In%20Adults%20With%20Major%20Depressive%20Disorder

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 898 potential participants were screened for this study. 804 participants were enrolled and received single-blind placebo during the screening period prior to randomization.
Groups:
- Placebo: Matching placebo tablets daily until Day 56 (Week 8) or early termination (ET).
- DVS SR 10 mg: Desvenlafaxine Succinate Sustained Release (DVS SR) 10 mg daily until Day 56 (Week 8) or ET.
- DVS SR 50 mg: DVS SR 50 mg daily until Day 56 (Week 8) or ET.
Period: Overall Study
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Started | 227 | 228 | 227
Treated | 223 | 226 | 224
Completed | 195 | 198 | 202
Not Completed | 32 | 30 | 25
Not completed — Adverse Event | 5 | 2 | 4
Not completed — Participant failed to return | 2 | 1 | 0
Not completed — Investigator request | 1 | 2 | 1
Not completed — Lack of Efficacy | 4 | 3 | 6
Not completed — Lost to Follow-up | 6 | 9 | 5
Not completed — Other | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 7 | 4
Not completed — Randomized not treated | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg | Total
Number analyzed (Participants) | 223 | 226 | 224 | 673
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.75 (12.85) | 41.01 (13.75) | 42.47 (13.47) | 41.74 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 135 | 135 | 409
  Male | 84 | 91 | 89 | 264
Hamilton Psychiatric Scale for Depression-17 item HAM-D17) total score [Mean (Standard Deviation); unit: Units on a scale] — HAM-D17 : a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
  Units on a scale | 23.23 (2.63) | 22.83 (2.26) | 23.12 (2.62) | 23.06 (2.51)
Clinical Global Impressions Scale-Severity of Illness (CGI-S) Score [Mean (Standard Deviation); unit: Units on a scale] — CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
  Units on a scale | 4.14 (0.35) | 4.14 (0.34) | 4.16 (0.39) | 4.14 (0.36)
Montgomery-Asberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: Units on a scale] — MADRS measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  Units on a scale | 28.33 (4.71) | 27.59 (4.49) | 28.44 (4.83) | 28.12 (4.69)
HAM-D6 total score [Mean (Standard Deviation); unit: Units on a scale] — HAM-D6: a standardized, clinician-administered rating scale that assesses 6 items associated with major depression and is a subset of the HAM-D17. HAM-D6 score ranges from 0-22. The scale uses HAM-D17 items: 1, 2, 7, 8, 10 and 13. Item 13 is scored 0-2 and all others are scored 0-4.
  Units on a scale | 12.72 (1.51) | 12.77 (1.41) | 12.63 (1.49) | 12.71 (1.47)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — SDS: a self-administered tool that measures functional impairment in 3 domains: Work/School, Social Life, and Family Life/Home Responsibilities.Participant rates extent to which each of these domains are impaired by his/her symptoms using 10 point visual analog scale:(0=not at all impaired,10=extremely impaired) for total maximum score of 30.
  Units on a scale | 16.88 (8.25) | 16.42 (8.37) | 17.06 (7.73) | 16.78 (8.12)
World Health Organization 5-Item Well-Being Index (WHO-5) [Mean (Standard Deviation); unit: Units on a scale] — WHO-5 evaluates positive psychological well-being. WHO-5 consists of 5 questions and each is rated on a 6-point scale. The total score ranges from 0 to 25 ( 0= worst possible quality of life; 25=best possible quality of life).
  Units on a scale | 7.39 (4.80) | 7.47 (4.86) | 7.06 (4.26) | 7.31 (4.65)
Participants with Sexual dysfunction [Number; unit: Percentage of Participants] — Arizona Sexual Experiences Scale (ASEX) includes 5 questions that evaluate sexual function exclusively during week prior to completion in the following areas: libido, excitability and ability to reach orgasm. Sexual dysfunction=ASEX total score of 19 or greater, or a score of 5 or greater on any item, or a score of 4 or greater on any 3 items.
  Percentage of Participants | 58.8 | 61.3 | 65.8 | 185.9
Participants with Columbia Suicide-Severity Rating Scale (C-SSRS) total score [Number; unit: Participants] — C-SSRS was mapped into Columbia Classification Algorithm of Suicide Assessment (C-CASA)(1-4) to prospectively assess whether participants experienced: completed suicide(1),suicide attempt(2),preparatory acts toward imminent suicidal behavior(3),suicidal ideation,any suicidal behavior and ideation(4).Participants with "yes" response were reported.
  Participants
    Completed Suicide | 0 | 0 | 0 | 0
    Suicide Attempt | 0 | 0 | 0 | 0
    Preparatory acts toward imminent suicidal behavior | 0 | 0 | 0 | 0
    Suicidal ideation | 37 | 31 | 29 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HAM-D17 Total Score at Final On-therapy (FOT) Evaluation (Week 8 or ET)
Description: HAM-D17: a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Baseline and Week 8 (or ET)
Population: Intent-To-Treat (ITT) Population:all randomly assigned participants with baseline primary efficacy evaluation, had taken at least 1 dose of double-blind drug and 1 primary efficacy evaluation after first dose of double-blind drug. If participant had missing value at any visit, last observation carried forward (LOCF) method of imputation was used.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Units on a scale | -8.42 (0.45) | -9.28 (0.45) | -8.92 (0.45)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; An analysis of covariance (ANCOVA) model with treatment and as a factor and the baseline HAM-D17 total score as a covariate was used to compare DVS SR 10 mg to placebo. The comparison was performed at the 0.05 level overall; Test type: Superiority or Other; p = 0.175, ANCOVA — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-0.38 to 2.10]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.421, ANCOVA — A Hochberg step-up procedure was used to control for the multiplicity associated with multiple active dose arms; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.73 to 1.75]

2. Secondary Outcome: Number of Participants With Categorical Scores on CGI-Improvement (CGI-I) at FOT Evaluation (Week 8 or ET)
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8 (or ET)
Population: ITT Population included all randomly assigned participants who had baseline primary efficacy evaluation, had taken at least 1 dose of double-blind study drug, and had at least 1 primary efficacy evaluation after first dose of double-blind study drug. If participant had a missing value at any visit, LOCF method of imputation was used.
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Participants
  1=Very much improved | 49 | 50 | 55
  2=Much improved | 54 | 75 | 53
  3=Minimally improved | 51 | 51 | 64
  4=No change | 61 | 46 | 49
  5=Minimally worse | 5 | 4 | 3
  6=Much worse | 3 | 0 | 0
  7=Very much worse | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Each DVS SR dose was separately compared to placebo. To control the study-wise type I error rate across the primary and the key secondary endpoints, as well as across the 2 active dose arms, testing of the key secondary hypothesis occurred only when both active doses were superior to placebo on the primary endpoint; Test type: Superiority or Other; p = 0.076, Cochran-Mantel-Haenszel — In this case, multiplicity arising from testing key secondary hypotheses in both doses was controlled by a Hochberg step-up procedure. p-Value obtained for the alternative hypothesis of 'Row mean scores differences'
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.204, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in Mean CGI-S Score at FOT Evaluation (Week 8 or ET)
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected.
Time Frame: Baseline and Week 8 (or ET )
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Units on a scale | -1.08 (0.07) | -1.23 (0.07) | -1.11 (0.07)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate; Test type: Superiority or Other; p = 0.130, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.04 to 0.35]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.757, ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.16 to 0.23]

4. Secondary Outcome: Change From Baseline in MADRS Total Score at FOT Evaluation (Week 8 or ET)
Description: MADRS measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline and Week 8 (or ET)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 222 | 224 | 222
Units on a scale | -9.87 (0.63) | -11.28 (0.63) | -10.76 (0.63)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.114, ANCOVA; Median Difference (Final Values) = 1.41, 95% CI 2-sided [-0.34 to 3.16]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.316, ANCOVA; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-0.85 to 2.64]

5. Secondary Outcome: Change From Baseline in HAM-D6 Total Score at FOT Evaluation (Week 8 or ET)
Description: HAM-D6: a standardized, clinician-administered rating scale that assesses 6 items characteristically associated with major depression and is a subset of HAM-D17. HAM-D6 score ranges from 0-22. 0=none/absent and 22=most severe.The scale uses HAM-D17 items: 1, 2, 7, 8, 10 and 13. Item 13 is scored 0-2 and all others are scored 0-4.
Time Frame: Baseline and Week 8 (or ET )
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Units on a scale | -4.75 (0.27) | -5.49 (0.27) | -5.19 (0.27)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.054, ANCOVA; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.01 to 1.50]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.253, ANCOVA; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.32 to 1.20]

6. Secondary Outcome: Number of Participants With a Response on the HAM-D17 at FOT Evaluation (Week 8 or ET)
Description: A HAM-D17 responder was defined as a participant with a 50% or greater decrease from baseline in HAM-D17 score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Week 8 (or ET)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Participants | 85 | 100 | 91
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using a logistic regression model with treatment as a factor and baseline HAM-D17 score as a covariate; Test type: Superiority or Other; p = 0.2415, Regression, Logistic; Odds Ratio (OR) = 1.254, 95% CI 2-sided [0.86 to 1.83]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.6169, Regression, Logistic; Odds Ratio (OR) = 1.102, 95% CI 2-sided [0.75 to 1.61]

7. Secondary Outcome: Number of Participants in Remission Based on the HAM-D17 at FOT Evaluation (Week 8 or ET)
Description: Remission was defined as a HAM-D17 score of less than or equal to 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Individual items are scored on either a 3 point (0 to 2) or a 5 point scale (0 to 4), with 0=none/absent and 4=most severe, for a maximum total score of 50.
Time Frame: Week 8 (or ET)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Participants | 42 | 52 | 39
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3667, Regression, Logistic; Odds Ratio (OR) = 1.236, 95% CI 2-sided [0.78 to 1.96]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.6509, Regression, Logistic; Odds Ratio (OR) = 0.894, 95% CI 2-sided [0.55 to 1.45]

8. Secondary Outcome: Number of Participants With a Response on the MADRS Score at FOT Evaluation (Week 8 or ET)
Description: A MADRS responder was defined as a participant with a 50% or greater decrease from baseline in MADRS score. It measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Week 8 (or ET)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 222 | 224 | 222
Participants | 84 | 95 | 90
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis would be conducted with a logistic regression model with treatment as a factor and baseline MADRS score as a covariate; Test type: Superiority or Other; p = 0.3893, Regression, Logistic; Odds Ratio (OR) = 1.182, 95% CI 2-sided [0.81 to 1.73]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.5510, Regression, Logistic; Odds Ratio (OR) = 1.123, 95% CI 2-sided [0.77 to 1.65]

9. Secondary Outcome: Number of Participants With a Response on the CGI-I Score at FOT Evaluation (Week 8 or ET)
Description: CGI-I responder was defined as a participant with a score of 1 (very much improved) or 2 (much improved) on the CGI-I. CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 8 (or ET)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Participants | 103 | 125 | 108
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis would be conducted with a logistic regression model with treatment as a factor; Test type: Superiority or Other; p = 0.0536, Regression, Logistic; Odds Ratio (OR) = 1.442, 95% CI 2-sided [0.99 to 2.09]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; Analysis would be conducted with a logistic regression model with treatment as a factor; Test type: Superiority or Other; p = 0.6679, Regression, Logistic; Odds Ratio (OR) = 1.085, 95% CI 2-sided [0.75 to 1.57]

10. Other Pre Specified Outcome: Population Pharmacokinetics for Desvenlafaxine Plasma Concentrations
Description: Relationship of demographic variables (age, gender, food, race, creatinine, aspartate aminotransaminase, alanine transaminase, bilirubin and concomitant medications) were examined by fitting measured DVS plasma concentrations to a 1 compartment model with first order absorption. Demographic variables were examined for clearance (CL/F), volume of distribution (V/F), Steady Area under Curve (AUC) using nonlinear mixed effects modeling. Final parameter estimates for demographic factors effecting CL/F, V/F and AUC were determined.
Time Frame: Week 2, 4 and 8 (or ET)
Population: PK population; data was insufficient examine the effect of demographic variables on the PK of desvenlafaxine. Parameter values were calculated for variables altering CL/F, AUC and V/F. Population parameters from nonlinear mixed effects modeling were not summarized as descriptive statistics.
Measure: Mean (Standard Deviation); unit: nanogram(ng)/mL
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Change From Baseline in SDS at FOT Evaluation (Week 8 or ET)
Description: SDS: a self-administered tools that measures functional impairment in 3 domains: Work/School, Social Life, and Family Life/Home Responsibilities. The participant rates the extent to which each of these domains is impaired by his/her symptoms using a 10 point visual analog scale: (0=not at all impaired, 10=extremely impaired) for a total maximum score of 30.
Time Frame: Baseline and Week 8 (or ET)
Population: ITT Population included all randomly assigned participants who had baseline primary efficacy evaluation,had taken at least 1 dose of double-blind study drug,had at least 1 primary efficacy evaluation after first dose of double-blind drug.'n' is participants who received drug and were evaluated for measure at timepoint for each group respectively.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Units on a scale
  Total Score (n=220,223,219) | -2.63 (0.48) | -4.09 (0.48) | -3.78 (0.49)
  Work/Studies Component(n=220,223,219) | -0.61 (0.17) | -1.10 (0.17) | -1.14 (0.17)
  Social Life and Leisure Activities(n=222,224,221) | -1.08 (0.18) | -1.58 (0.17) | -1.36 (0.18)
  Family Life/Home Responsibilities (n=222,224,221) | -0.98 (0.17) | -1.43 (0.17) | -1.20 (0.17)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for "total score"; Test type: Superiority or Other; p = 0.033, ANCOVA; Mean Difference (Final Values) = 1.46, 95% CI 2-sided [0.12 to 2.79]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.096, ANCOVA; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-0.20 to 2.49]
Statistical Analysis 3: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for "work/studies component score"; Test type: Superiority or Other; p = 0.043, ANCOVA; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.02 to 0.95]
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.027, ANCOVA; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [0.06 to 1.00]
Statistical Analysis 5: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for "social life and leisure activities component score"; Test type: Superiority or Other; p = 0.045, ANCOVA; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [0.01 to 0.98]
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p = 0.277, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.22 to 0.76]
Statistical Analysis 7: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using ANCOVA on the change from baseline with treatment as a factor and corresponding baseline value as a covariate for "family life/home responsibilities component score"; Test type: Superiority or Other; p = 0.056, ANCOVA; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.01 to 0.91]
Statistical Analysis 8: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.355, ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.24 to 0.68]

12. Other Pre Specified Outcome: Change From Baseline in WHO-5 Total Score at FOT Evaluation (Week 8 or ET)
Description: WHO-5 evaluates positive psychological well-being. WHO-5 consists of 5 questions and each is rated on a 6-point scale. The total score ranges from 0 to 25 (0= worst possible quality of life; 25=best possible quality of life).
Time Frame: Baseline and Week 8 (or ET)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 222 | 224 | 221
Units on a scale | 2.96 (0.36) | 4.51 (0.35) | 3.73 (0.36)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-2.53 to -0.56]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.129, ANCOVA; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.75 to 0.22]

13. Other Pre Specified Outcome: Percentage of Participants With Sexual Dysfunction at FOT Evaluation (Week 8 or ET)
Description: ASEX scale includes 5 questions that evaluate sexual function exclusively during the week prior to completion in the following areas: libido, excitability and ability to reach orgasm. Sexual dysfunction=an ASEX total score of 19 or greater, or a score of 5 or greater on any item, or a score of 4 or greater on any 3 items. Participants who have had no sexual activity during the prior week were instructed to not complete questions 3 through 5.
Time Frame: Week 8 (or ET)
Population: The safety population included all participants randomly assigned to treatment who had taken at least 1 dose of double-blind study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 221 | 222 | 220
Percentage of Participants | 52.0 | 48.6 | 59.5
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; Analysis was conducted using a logistic regression model with treatment and gender as factors and baseline sexual dysfunction status as a covariate; Test type: Superiority or Other; p = 0.3097, Regression, Linear; Odds Ratio (OR) = 0.800, 95% CI 2-sided [0.52 to 1.23]
Statistical Analysis 2: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.2794, Regression, Logistic; Odds Ratio (OR) = 1.272, 95% CI 2-sided [0.82 to 1.97]

14. Other Pre Specified Outcome: Number of Participants With Categorical Scores on the C-SSRS at FOT Evaluation (Week 8 or ET)
Description: C-SSRS mapped into C-CASA(1-7) to assess whether participant:completed suicide(1),suicide attempt(2)(response of "Yes" on "Actual Attempt"),preparatory acts toward imminent suicidal behavior (3)("Yes" on "Preparatory Acts or Behavior"),suicidal ideation (4)("Yes" on "Wish to be dead","Non-Specific Active Suicidal Thoughts","Active Suicidal Ideation with methods without Intent to Act or Some Intent to Act,without Specific Plan or with Specific Plan and Intent),any suicidal behavior or ideation,self-injurious behaviour(7)("Yes" on "Has subject engaged in Non-suicidal Self-Injurious Behavior").
Time Frame: Week 8 (or ET)
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Participants
  Completed suicide | 0 | 0 | 0
  Suicide attempt | 0 | 1 | 0
  Preparatory acts toward imminent suicidal behavior | 0 | 0 | 1
  Suicidal ideation | 56 | 43 | 45
  Any suicidal behavior and/or ideation | 56 | 43 | 45
  Self-injurious behavior, no suicidal intent | 1 | 0 | 0

15. Other Pre Specified Outcome: Discontinuation-Emergent Signs and Symptoms (DESS)
Description: DESS: a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article. The DESS total score is the sum of the number of new symptoms and old (but worse) symptoms that appeared during tapering of the test article. A higher score indicates more symptoms.
Time Frame: Week 8 to 10 (or ET)
Population: Analysis included completers for exposure (those whose exposure duration was at least 53 days) among safety population. 'n' is participants who received drug and were evaluated for measure at timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Number analyzed (Participants) | 223 | 226 | 224
Units on a scale
  Week 8 (or ET) (n=190,194,191) | 0.72 (1.81) | 0.80 (1.78) | 0.83 (2.05)
  Week 9 ( or ET + 1 week) (n=178,185,186) | 1.26 (2.78) | 1.08 (2.31) | 1.98 (3.29)
  Week 10 (or ET + 2 weeks (n=170,182,182) | 0.90 (2.30) | 0.91 (2.24) | 1.07 (2.50)
Statistical Analysis 1: Comparison: Placebo vs DVS SR 10 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate was used at Week 8; Test type: Superiority or Other; p = 0.805, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs DVS SR 10 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate was used at Week 9; Test type: Superiority or Other; p = 0.805, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs DVS SR 10 mg; To address the multiplicity effect inherent in these comparisons, adjusted p-values based on the false discovery rate was used at Week 10; Test type: Superiority or Other; p = 0.978, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.805, Regression, Logistic
Statistical Analysis 5: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.154, t-test, 2 sided
Statistical Analysis 6: Comparison: Placebo vs DVS SR 50 mg; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.805, t-test, 2 sided

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | DVS SR 10 mg | DVS SR 50 mg
Serious Adverse Events (participants affected / at risk) | 3/223 | 1/226 | 1/224
Other Adverse Events (participants affected / at risk) | 166/223 | 168/226 | 170/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | DVS SR 10 mg (N=226) | DVS SR 50 mg (N=224)
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | DVS SR 10 mg (N=226) | DVS SR 50 mg (N=224)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 2 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 5 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 1 | 4
Ventricular extrasystoles (Cardiac disorders) | 2 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 2
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Blepharospasm (Eye disorders) | 2 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 3
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 1
Excessive eye blinking (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 2 | 2 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Miosis (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 1
Photopsia (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 3 | 3 | 4
Visual impairment (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 3
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 8 | 15
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 20 | 19
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 13 | 20 | 25
Dyspepsia (Gastrointestinal disorders) | 7 | 6 | 9
Eructation (Gastrointestinal disorders) | 0 | 3 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 7 | 5 | 2
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 21 | 26 | 42
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 5
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 9 | 6
Vomiting in pregnancy (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 2 | 0 | 2
Fatigue (General disorders) | 8 | 10 | 16
Feeling abnormal (General disorders) | 0 | 0 | 1
Feeling jittery (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 2 | 4
Injection site pruritus (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 12 | 8 | 8
Non-cardiac chest pain (General disorders) | 0 | 1 | 3
Oedema peripheral (General disorders) | 1 | 2 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 4
Temperature intolerance (General disorders) | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 3
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 4 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 4 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 1
Infected bites (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 7 | 8 | 5
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5 | 7
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 3 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 2
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 1 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 17 | 21 | 16
Urinary tract infection (Infections and infestations) | 4 | 1 | 1
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 4 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 2 | 1 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Blood human chorionic gonadotropin (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 2 | 0
Blood pressure diastolic decreased (Investigations) | 1 | 1 | 1
Blood pressure diastolic increased (Investigations) | 1 | 2 | 0
Blood pressure increased (Investigations) | 0 | 1 | 4
Blood pressure orthostatic decreased (Investigations) | 0 | 1 | 0
Blood pressure systolic decreased (Investigations) | 0 | 1 | 0
Blood prolactin increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 2 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 3 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Platelet count increased (Investigations) | 0 | 1 | 0
Protein urine (Investigations) | 0 | 1 | 0
Tuberculin test positive (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 3 | 1 | 1
Weight increased (Investigations) | 2 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 0
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 10 | 20
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Food craving (Metabolism and nutrition disorders) | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 6
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Crying (Nervous system disorders) | 2 | 1 | 3
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 7 | 3
Dizziness (Nervous system disorders) | 17 | 11 | 29
Dizziness postural (Nervous system disorders) | 1 | 2 | 5
Drug withdrawal headache (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Dyskinesia (Nervous system disorders) | 0 | 1 | 0
Exaggerated startle response (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 23 | 32 | 24
Hypersomnia (Nervous system disorders) | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Hypogeusia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 1 | 1
Migraine (Nervous system disorders) | 2 | 0 | 3
Paraesthesia (Nervous system disorders) | 4 | 3 | 5
Poor quality sleep (Nervous system disorders) | 1 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 3 | 1 | 1
Sedation (Nervous system disorders) | 1 | 1 | 1
Sinus headache (Nervous system disorders) | 1 | 1 | 4
Somnolence (Nervous system disorders) | 12 | 10 | 13
Syncop (Nervous system disorders) | 0 | 0 | 1
Tension headache (Nervous system disorders) | 8 | 7 | 11
Tremor (Nervous system disorders) | 5 | 3 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1
Abnormal dreams (Psychiatric disorders) | 8 | 11 | 14
Agitation (Psychiatric disorders) | 0 | 0 | 2
Anger (Psychiatric disorders) | 0 | 1 | 2
Anorgasmia (Psychiatric disorders) | 0 | 2 | 3
Anxiety (Psychiatric disorders) | 6 | 7 | 7
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 1
Bruxism (Psychiatric disorders) | 1 | 2 | 0
Depersonalisation (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 8 | 0
Derealisation (Psychiatric disorders) | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Dissociation (Psychiatric disorders) | 2 | 3 | 1
Distractibility (Psychiatric disorders) | 0 | 1 | 0
Elevated mood (Psychiatric disorders) | 2 | 0 | 0
Impulse-control disorder (Psychiatric disorders) | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 2 | 1 | 5
Insomnia (Psychiatric disorders) | 14 | 16 | 20
Libido decreased (Psychiatric disorders) | 5 | 5 | 6
Loss of libido (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 2 | 0 | 0
Middle insomnia (Psychiatric disorders) | 1 | 5 | 5
Mood altered (Psychiatric disorders) | 0 | 2 | 3
Mood swings (Psychiatric disorders) | 1 | 1 | 2
Nervousness (Psychiatric disorders) | 0 | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 6 | 4
Orgasm abnormal (Psychiatric disorders) | 1 | 2 | 2
Orgasmic sensation decreased (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 3 | 0
Panic disorder (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 2
Self injurious behaviour (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 5 | 3 | 6
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Tearfulness (Psychiatric disorders) | 1 | 3 | 4
Terminal insomnia (Psychiatric disorders) | 2 | 0 | 3
Withdrawal syndrome (Psychiatric disorders) | 8 | 12 | 16
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2
Urge incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 4
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 2 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Ejaculation delayed (Reproductive system and breast disorders) | 1 | 2 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 | 3
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 2
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 11 | 12
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 6 | 3 | 4
Hypertension (Vascular disorders) | 4 | 0 | 2
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.